CLINICAL TRIAL: NCT00708474
Title: OsseoFit™ Porous Tissue Matrix™ Prospective Data Collection
Brief Title: OsseoFit™ Prospective Data Collection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Planning new study protocol
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSM2008001
Record Dates: First submitted 2008-06-25; First posted 2008-07-02 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Bone Graft; Knee
Keywords: Bone graft; Bone void filler; Bone plug; OsseoFit™; knee; bone graft sites in the knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OsseoFit™ (Experimental): Treatment of bone graft site with OsseoFit™ Porous Tissue Matrix™.
  Interventions: Device: OsseoFit™ Porous Tissue Matrix™
- Open (No Intervention): Treatment of bone graft site without OsseoFit™ Porous Tissue Matrix™.

INTERVENTIONS:
Device: OsseoFit™ Porous Tissue Matrix™ — Bone void filler
  Arms: OsseoFit™

SUMMARY:
This study compares the fill of bone graft sites in the knee. It is hypothesized that harvest sites, voids, and defects caused by trauma that are treated with the OsseoFit™ Porous Tissue Matrix™ device will achieve a better fill grade than those treated with the conventional method.

ELIGIBILITY:
Inclusion Criteria:

* The OsseoFit™ Porous Tissue Matrix™ is intended to be gently packed into the bony voids or gaps of the extremities and pelvis caused by trauma or surgery and are not intrinsic to the stability of the bony structure. These defects may be created from repetitive motion or traumatic injury to the bone or surgically created osseous defects for the harvest of bone. The device is a bone void filler that resorbs and is replaced with bone during the healing process. The device may be combined with sterile fluids such as saline or autogenous blood products such as blood, platelets, or bone marrow aspirate. The addition of these autogenous blood products does not compromise the performance of the device. Hydration with biologically beneficial sterile fluids can potentially have a positive influence on the healing and replacement of the device with bone.

Exclusion Criteria:

* Infection at site
* Hypercalcemia
* Known allergies to bovine collagen
* Current osteomyelitis at operative site
* Systemic conditions which affect bone and/or wound healing
* Known severe allergies manifested by history of anaphylaxis
* Desensitization treatment injections to meat products, as injections may contain bovine collagen
* Severe degenerative bone disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Site repair grade by MRI analysis | 6 months

SECONDARY OUTCOMES:
Site repair grade by MRI analysis | 3 months, 1 year
Pain Score | 3 months, 6 months, 1 year
Function Score | 3 months, 6 months, 1 year
Physical Evaluation | 3 months, 6 months, 1 year
Incidence of adverse events | Any time

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Lehman, M.D., Principal Investigator
Locations (1):
- Biomet Sports Medicine, Warsaw, Indiana, United States